CLINICAL TRIAL: NCT01981031
Title: Phase 1 Study to Assess the Efficacy and Safety of BioChaperone® Combo and Humalog® Mix 25 in Subjects With Type 1 Diabetes
Brief Title: A Trial to Assess the Efficacy and Safety of BioChaperone Combo and Humalog Mix 25 in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BC3-CT005
Record Dates: First submitted 2013-10-31; First posted 2013-11-11 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2014-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Drug: BioChaperone® Combo
  Interventions: Drug: BioChaperone® Combo
- B (Active Comparator): Drug: Humalog® Mix25
  Interventions: Drug: Humalog® Mix25

INTERVENTIONS:
Drug: BioChaperone® Combo — Single dose of 0.8U/kg body weight injected subcutaneously (under the skin)
  Arms: A
Drug: Humalog® Mix25 — Single dose of 0.8U/kg body weight injected subcutaneously (under the skin)
  Arms: B

SUMMARY:
BioChaperone Combo is a liquid formulation containing both Insulin Glargine and Insulin Lispro.

The aim of this trial is to assess the efficacy and safety of BioChaperone® Combo in subjects with type 1 diabetes under a dose of 0.8 U/kg.

This trial is a phase 1 single-center, randomized, double-blinded, two-treatment, two-period cross-over, 30-hour euglycaemic glucose clamp trial in subjects with type 1 diabetes mellitus. Each subject will be randomly allocated to one single dose of 0.8 U/kg of BioChaperone® Combo and to one single dose of 0.8 U/kg of Humalog® Mix 25 on two separate dosing visits.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least (or equal to ) 12 months,
* Treated with multiple daily insulin injections or insulin pump treatment for at least (or equal to) 12 months,
* Body Mass Index (BMI): 18.0-28.0kg/m2 (both inclusive)

Exclusion Criteria:

* Type 2 diabetes mellitus,
* The receipt of any investigational product within 3 month prior to first dosing,
* Clinically significant abnormalities, as judged by the investigator,
* Any systemic treatment with drugs known to interfere with glucose metabolism,
* History of alcoholism or drug/chemical abuse and any tobacco product within 5 years prior to screening
* Blood or plasma donation in the past month or more than 500mL within 3 months prior to screening

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
End of action of 0.8 U/kg BioChaperone® Combo (time from administration until blood glucose concentration is consistently above 8.3 mmol/L during the glucose clamp procedure) | from 0 to 30 hours after a single-dose administration

SECONDARY OUTCOMES:
Compare pharmacodynamics and pharmacokinetics profiles between BioChaperone® Combo and Humalog® Mix25 | from 0 to 30 hours after a single-dose administration
Number of Adverse Events | Weeks 0-10
  hypoglycemic events, local tolerability, adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Neuss, Germany